CLINICAL TRIAL: NCT00232427
Title: Optimized Therapy of Decompensated Liver Cirrhosis by Hemodynamic Monitoring Using the PiCCO System
Brief Title: PiCCO Guided Therapy in Liver Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PiCCO
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2007-10-03 (Estimated); Status verified 2007-09

CONDITIONS: Liver Cirrhosis
Keywords: Liver cirrhosis; Hemodynamics; Fluid balance
MeSH Terms: conditions — Liver Cirrhosis

INTERVENTIONS:
Procedure: Hemodynamic monitoring system PiCCO

SUMMARY:
Prospective comparison of standard therapy in liver cirrhosis versus standard therapy plus intensified hemodynamic monitoring using the PiCCO system.

DETAILED DESCRIPTION:
Patients presenting with advanced liver cirrhosis will receive either standard treatment or standard treatment plus hemodynamic monitoring with the PiCCO device. Fluids and vasoacitve drugs will be administered according to the measurements over a period of 5 days.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis Child-Pugh-Score > 7
* Ascites > 500 ml

Exclusion Criteria:

* Coronary heart disease
* Apoplexia < 6 months ago
* Vasculitis
* Thrombosis
* Arterial occlusive disease > stadium II

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-08; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Survival

SECONDARY OUTCOMES:
Renal complications
Length of intensive care
Change in APACHE II

CONTACTS AND LOCATIONS:
Overall Officials: Jens Encke, PD Dr. med., Principal Investigator — Heidelberg University
Locations (1):
- University of Heidelberg, Clinical center, Heidelberg, Germany